CLINICAL TRIAL: NCT02638220
Title: An Observational, Multicenter Study of the Prevalence of Cerebrotendinous Xanthomatosis (CTX) in Patient Populations Diagnosed With Early-Onset Idiopathic Bilateral Cataracts
Brief Title: Cerebrotendinous Xanthomatosis (CTX) Prevalence Study
Status: Completed | Type: Observational
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 018CTXX15001
Record Dates: First submitted 2015-11-23; First posted 2015-12-23 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: Cerebrotendinous Xanthomatosis (CTX)
Keywords: Cerebrotendinous Xanthomatosis; CTX Prevalence Study; CTX; Idiopathic Bilateral Cataracts; Cataracts; Bilateral Cataracts; Early-Onset Idiopathic Bilateral Cataracts; Observational Study; Ophthalmology
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Iiopathic bilateral cataracts occur in many children with Cerebrotendinous Xanthomatosis (CTX) so the opportunity to use contact with health care providers in connection with pediatric cataract evaluation and treatment is a promising avenue for disease detection and prevention.

DETAILED DESCRIPTION:
This is an observational, multicenter study to determine the prevalence of Cerebrotendinous Xanthomatosis (CTX) in patient populations diagnosed with early-onset idiopathic bilateral cataracts. Patients who are potentially eligible for study participation will be identified through a chart review of patients who were seen at each study site prior to that site's initiation, or by entering care at the site while the site is participating in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of idiopathic bilateral cataracts
2. Between the ages of 2 to 21 years at the time of diagnosis

Exclusion Criteria:

1. The patient has a diagnosis of cataracts with known etiology other than CTX
2. The patient has a diagnosis of CTX
3. The patient has cataracts caused by cataractogenic treatments
4. The patient has taken or is currently taking cholic acid or chenodeoxycholic acid
5. The patient has participated in an interventional clinical trial in the past 30 days
6. The patient and/or their parent/legal guardian, in the opinion of the Investigator, is unable to adhere to the requirements of the study

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Early-Onset Idiopathic Bilateral Cataracts
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2015-09; Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Clinical Development Nephrology, Study Director — Travere Therapeutics, Inc.
Locations (41):
- United States (41):
  - Travere Investigational Site, Birmingham, Alabama
  - Travere Investigational Site, La Jolla, California
  - Travere Investigational Site, Los Angeles, California
  - Travere Investigational Site, Palo Alto, California
  - Travere Investigational Site, Aurora, Colorado
  - Travere Investigational Site, Gainesville, Florida
  - Travere Investigational Site, Jacksonville, Florida
  - Travere Investigational Site, Atlanta, Georgia
  - Travere Investigational Site, Chicago, Illinois
  - Travere Investigational Site, Indianapolis, Indiana
  - Travere Investigational Site, Iowa City, Iowa
  - Travere Investigational Site, Louisville, Kentucky
  - Travere Investigational Site, New Orleans, Louisiana
  - Travere Investigational Site, Baltimore, Maryland
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site, Ann Arbor, Michigan
  - Travere Investigational Site, Detroit, Michigan
  - Travere Investigational Site, Kansas City, Missouri
  - Travere Investigational Site, St Louis, Missouri
  - Travere Investigational Site, The Bronx, New York
  - Travere Investigational Site, Chapel Hill, North Carolina
  - Travere Investigational Site, Durham, North Carolina
  - Travere Investigational Site, Cincinnati, Ohio
  - Travere Investigational Site, Cleveland, Ohio
  - Travere Investigational Site, Columbus, Ohio
  - Travere Investigational Site, Oklahoma City, Oklahoma
  - Travere Investigational Site, Portland, Oregon
  - Travere Investigational Site, Tigard, Oregon
  - Travere Investigational Site, Philadelphia, Pennsylvania
  - Travere Investigational Site, Charleston, South Carolina
  - Travere Investigational Site, Germantown, Tennessee
  - Travere Investigational Site, Nashville, Tennessee
  - Travere Investigational Site, Houston, Texas
  - Travere Investigational Site, Salt Lake City, Utah
  - Travere Investigational Site, Norfolk, Virginia
  - Travere Investigational Site, Richmond, Virginia
  - Travere Investigational Site, Seattle, Washington
  - Travere Investigational Site, Spokane, Washington
  - Travere Investigational Site, Tacoma, Washington
  - Travere Investigational Site, Morgantown, West Virginia
  - Travere Investigational Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from 05 November 2015 through study completion on 19 February 2021.There were 43 sites in the United States included in the study.
Groups:
- Participants With CTX: Patients must have been between the ages of 2 and 21 at the time of diagnosis with idiopathic bilateral cataracts. Patients were excluded from the study if they had a diagnosis of cataracts with known etiology other than CTX, had cataracts caused by cataractogenic treatments, or the patient was taking cholic acid or chenodeoxycholic acid.
Period: Overall Study
Arm/Group | Participants With CTX
Started | 442
Completed | 426
Not Completed | 16
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Withdrawn, sample error, non-adherence, illness | 6

BASELINE CHARACTERISTICS:
Groups:
- Observational: Patients must have been between the ages of 2 and 21 at the time of diagnosis with idiopathic bilateral cataracts. Patients were excluded from the study if they had a diagnosis of cataracts with known etiology other than CTX, had cataracts caused by cataractogenic treatments, or the patient was taking cholic acid or chenodeoxycholic acid.
Arm/Group | Observational
Number analyzed (Participants) | 442
Age, Continuous [Mean (Full Range); unit: years] | 11.1 [0.1 to 52.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71
  Not Hispanic or Latino | 340
  Unknown or Not Reported | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 62
  White | 296
  More than one race | 22
  Unknown or Not Reported | 41
Region of Enrollment [Number; unit: participants]
  United States | 442

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Positive Genetic Test Results
Description: genetic test results
Time Frame: At genetic testing
Measure: Number; unit: Participants
Groups:
- Participants With CTX: Participants with bilateral cataracts and CTX
Arm/Group | Participants With CTX
Number analyzed (Participants) | 442
Participants | 4

ADVERSE EVENTS:
Time Frame: 4 hours
Description: Only Serious Adverse Events (SAEs) that were related to a research procedure (eg, blood sample collection) were to be recorded.
Arm/Group | Observational
All-Cause Mortality (participants affected / at risk) | 0/442
Serious Adverse Events (participants affected / at risk) | 0/442
Other Adverse Events (participants affected / at risk) | 0/442

LIMITATIONS AND CAVEATS:
This was an observational study; no treatment was administered and therefore no efficacy assessment was conducted. The results presented are used to evaluate the prevalence of CTX in a patient population diagnosed with early-onset idiopathic bilateral cataracts.

Only SAEs that were related to a research procedure (eg, blood sample collection) were to be recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02638220/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02638220/SAP_001.pdf